CLINICAL TRIAL: NCT07256171
Title: Cholesterol Optimization After Stroke: a Multicenter Prospective Study on LDL Cholesterol Control in Patients With Acute Stroke.
Brief Title: COAST Study - Cholesterol Optimization After Stroke
Acronym: COAST
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Frisullo Giovanni, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 8247
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Stroke (CVA) or Transient Ischemic Attack; Cerebral Hemorrhage
Keywords: LDL cholesterol; lipid-lowering agents; statins; ezetimibe; bempedoic acid; PCSK9 inhibitors; stroke; cerebral hemorrhage; transient ischemic attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Cerebral Hemorrhage | interventions — Diet, Fat-Restricted; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; PCSK9 Inhibitors; Fibric Acids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: low-fat diet, supplements, statins, ezetimibe, bempedoic acid, PCSK9 inhibitors, fibrates, or other lipid-lowering agents — Low-Fat Diet Typical components: Increased fruits, vegetables, whole grains, lean proteins, and limited fried or processed foods.
  Supplements Non-prescription substances that can help reduce cholesterol, often used alongside diet or drugs. Plant sterols/stanols: Reduce cholesterol absorption in the intestine.
  Statins The first-line pharmacological treatment for high cholesterol. Mechanism: Inhibit HMG-CoA reductase, the key enzyme in cholesterol synthesis in the liver.
  Ezetimibe A cholesterol absorption inhibitor. Mechanism: Blocks intestinal absorption of dietary and biliary cholesterol.
  Bempedoic Acid A newer oral lipid-lowering drug. Mechanism: Inhibits ATP-citrate lyase, an enzyme upstream of HMG-CoA reductase in the cholesterol synthesis pathway.
  PCSK9 Inhibitors Monoclonal antibodies or siRNA therapies given by injection every 2-4 weeks (or biannually for inclisiran).
  Fibrates Drugs that primarily lower triglycerides and can modestly raise HDL cholesterol.

SUMMARY:
This study (acronym COAST Trial) is a multicenter observational registry aiming to document: patients' adherence and persistence to lipid-lowering therapy prescribed for secondary prevention; the proportion of patients achieving LDL cholesterol therapeutic targets at 3 months; the incidence of cerebrovascular recurrence and mortality at 90 days, as well as the occurrence of any adverse effects from these therapies. This information will provide a snapshot of post-stroke/TIA lipid-lowering management across centers and identify areas for improvement, offering useful data to optimize secondary prevention strategies in everyday clinical practice.

DETAILED DESCRIPTION:
SYNOPSIS STUDY TITLE COAST Study - Cholesterol Optimization After Stroke: a multicenter prospective study on LDL cholesterol control in patients with acute stroke.

ACRONYM COAST (COAST - Cholesterol Optimization After Stroke Trial: a multicenter prospective study on LDL cholesterol control in patients with acute stroke) SPONSOR Agostino Gemelli University Hospital Foundation IRCCS L.go Francesco Vito 1, 00168 Rome CRO N/A CO-FUNDER N/A PRINCIPAL INVESTIGATOR Dr. Giovanni Frisullo Head, UOSD Emergency Neurology BACKGROUND AND RATIONALE OF THE STUDY Stroke is the leading cause of disability and among the main causes of mortality worldwide. A significant proportion of patients with stroke have large-vessel atherosclerosis or other vascular risk factors; therefore, aggressive management of plasma lipids is crucial for secondary prevention. In routine clinical practice, the assessment of the lipid profile and the control of hypercholesterolemia are extremely variable, encompassing low-fat diets, various supplements, or medications. In light of these considerations, a prospective real-life study is needed to evaluate how patients with ischemic stroke, hemorrhagic stroke, or TIA are managed regarding lipid profile assessment and LDL-C control in secondary prevention. This study (acronym COAST Trial) is a multicenter observational registry aiming to document: patients' adherence and persistence to lipid-lowering therapy prescribed for secondary prevention; the proportion of patients achieving LDL cholesterol therapeutic targets at 3 months; the incidence of cerebrovascular recurrence and mortality at 90 days, as well as the occurrence of any adverse effects from these therapies. This information will provide a snapshot of post-stroke/TIA lipid-lowering management across centers and identify areas for improvement, offering useful data to optimize secondary prevention strategies in everyday clinical practice.

STUDY OBJECTIVES

Primary:

To assess patients' adherence and persistence to lipid-lowering therapy prescribed for secondary prevention (low-fat diet, supplements, statins, ezetimibe, bempedoic acid, PCSK9 inhibitors, fibrates, or other lipid-lowering agents) 3 months after the acute cerebrovascular event (ischemic stroke, intracerebral hemorrhage, or TIA).

Secondary:

Lipid target attainment: determine the proportion of patients who, at 90 ± 15 days from the acute event, achieve the pre-specified LDL cholesterol goals (e.g., <55 mg/dL for ischemic stroke patients, <40 mg/dL for patients already on intensive lipid-lowering therapy, etc.).

Recurrence of cerebrovascular events: record the incidence of new cerebrovascular events within 90 ± 15 days of the index event, including recurrent ischemic stroke, hemorrhagic stroke, or TIA. This objective considers a composite endpoint of cerebrovascular recurrence; the incidence of each event type (ischemic stroke, hemorrhagic stroke, TIA) will also be assessed separately.

Occurrence of cardiovascular events: record the incidence of cardiovascular events (acute myocardial infarction, unstable angina, critical coronary artery disease) attributable to atherosclerotic disease within 90 ± 15 days of the index event.

Mortality: monitor all-cause mortality within 90 ± 15 days and distinguish the proportion of deaths attributable to cerebrovascular causes (e.g., fatal stroke) versus other causes.

Safety of lipid-lowering therapy: assess the frequency of adverse events potentially related to lipid-lowering therapy during the 90 ± 15-day follow-up (e.g., muscle events such as myalgias or myopathies, elevation of liver enzymes, onset of diabetes, injection-site reactions for agents such as PCSK9 inhibitors, etc.) and verify whether therapy suspension or modification is required due to such events.

Monitoring of laboratory parameters: monitor the evolution of key laboratory parameters from baseline to 90 ± 15 days, with particular attention to the lipid profile (LDL, HDL, total cholesterol, triglycerides), and other relevant tests (e.g., glucose/HbA1c, renal function, liver function via ALT/AST, C-reactive protein, Lp(a)), to assess metabolic response to lipid-lowering treatment and identify any significant alterations (e.g., transaminase increases).

Functional disability: optionally, assess global functional outcome at 90 ± 15 days using the mRS (modified Rankin Scale) score, if collected during follow-up, to provide an indication of the patient's overall neurological status.

ENDPOINTS

Primary:

Adherence to lipid-lowering therapy, defined as the percentage of patients who are adherent (intake of ≥80% of prescribed doses) and persistent (on therapy without interruptions) at the end of follow-up. Rates of persistence (patients who did not discontinue therapy) and adherence (patients who took it regularly) may also be considered separately.

Secondary:

Proportion of patients achieving an LDL target value (for example, <55 mg/dL for ischemic stroke patients, <40 mg/dL for patients already on maximal therapy, etc.) at the 90 ± 15-day follow-up. This endpoint reflects the overall effectiveness of lipid-lowering management in bringing patients to the recommended target.

Recurrence of stroke (ischemic or hemorrhagic), TIA, or acute cardiovascular events (myocardial infarction or angina) within 90 ± 15 days of the index event (composite endpoint). The incidence of recurrent ischemic stroke, hemorrhagic stroke, and TIA will also be analyzed separately as secondary individual endpoints.

All-cause mortality at 90 ± 15 days. In parallel, cerebrovascular mortality (deaths attributable to the direct consequences of stroke or other cerebrovascular events) will be analyzed relative to mortality from other causes.

Change in lipid levels and other laboratory parameters from baseline to 90 ± 15 days. In particular, change in LDL (continuous, in mg/dL) will be a secondary endpoint measuring response to therapy; mean changes in total cholesterol, HDL, triglycerides, as well as any variation in ALT/AST, HbA1c, and other available markers will be assessed to monitor efficacy and metabolic safety.

Adverse events related to lipid-lowering medications: incidence of clinically relevant side effects reported within 90 ± 15 days (e.g., myalgias without significant CK elevation, gastrointestinal disturbances from fibrates, injection-site reactions with PCSK9 inhibitors, etc.). These will contribute to the overall evaluation of therapy tolerability.

Functional disability at 90 ± 15 days: optionally assessed using the mRS (modified Rankin Scale) score if captured at follow-up, to provide an overview of overall clinical outcome.

STUDY DESIGN Prospective observational study with medicinal products, multicenter. NUMBER OF PATIENTS 500 total patients. TARGET POPULATION Patients will be included with any etiological subtype of ischemic stroke (e.g., cardioembolic, atherosclerotic, lacunar, etc.) or hemorrhagic stroke or TIA.

INCLUSION CRITERIA

Inclusion criteria: All subjects meeting all of the following criteria at the time of enrollment will be included:

* Age ≥ 18 years, both sexes.
* Recent acute cerebrovascular event, defined as a confirmed diagnosis of ischemic stroke, hemorrhagic stroke, or TIA occurring less than 30 days prior to enrollment.
* Availability of a baseline measured LDL cholesterol value (direct or calculated) at the time of the index event or close to it.
* Patients for whom, in routine clinical practice, a lipid-lowering therapy has been indicated and prescribed for secondary prevention (low-fat diet, supplements, statins, ezetimibe, bempedoic acid, PCSK9 inhibitors, fibrates, or other lipid-lowering agents).
* Written informed consent obtained and signed by the patient before inclusion. If the patient is unable to provide consent autonomously (e.g., due to aphasia, impaired consciousness, etc.), informed consent will be obtained from a legal representative or proxy, in accordance with applicable regulations.

EXCLUSION CRITERIA

Exclusion criteria: Subjects presenting at least one of the following conditions will be excluded:

* Comorbidities or conditions preventing 3-month follow-up: e.g., terminal oncological disease with life expectancy <3 months, severe cognitive impairment (e.g., advanced dementia), or other conditions that make it impossible to obtain follow-up information; inability to contact the patient after discharge (e.g., non-resident foreign patient or lacking telephone contacts).
* Any other clinical, psychological, or social condition that, in the investigator's judgment, may compromise the patient's ability to adhere to the study or the reliability of the collected data.

STUDY DURATION AND ENROLLMENT PERIOD Each enrolled patient will be followed for 90 days; therefore, the last follow-up visit will occur approximately 3 months after the inclusion of the last patient. Considering possible delays, the total project duration (from initiation to last visit) is approximately 12 months. An interim analysis will be performed about 4 months after study start.

Enrollment duration: 6 months Follow-up duration: 3 months Total study duration: 12 months VARIABLES AND DATA COLLECTION The study foresees the collection of demographic, clinical, laboratory, instrumental data, and details of the treatments administered.

Specifically, at the follow-up visit (which may also be conducted by telephone), performed according to routine clinical practice at 3 months ± 2 weeks, the following parameters will be collected:

* Patient's clinical status (mRS, any new cerebrovascular events, adverse events, other…)
* Medication history
* Any laboratory tests including lipid profile For specifics, refer to the protocol. Data will be collected from patients' medical records. SAFETY/REGULATORY MANAGEMENT OF ADVERSE EVENTS All adverse events will be collected, recorded, and assessed for severity and relationship to the medicinal products under study and others, for the purpose of identifying suspected adverse reactions.

Every suspected adverse reaction will be reported to the National Competent Authority (AIFA), regardless of severity, according to the post-marketing pharmacovigilance process provided by the Ministerial Decree of April 30, 2015 and GVP (Good Pharmacovigilance Practices) Module VI, by notifying the Local Pharmacovigilance Officer for entry into the National Pharmacovigilance Network and, where required, the Ethics Committee.

SAFETY REFERENCE DOCUMENT SmPC (Summary of Product Characteristics). STATISTICAL ANALYSIS AND SAMPLE SIZE As this is not an interventional superiority study with predefined hypotheses, the statistical analysis will mainly be descriptive, aimed at quantifying outcome parameters and exploring associations with patient characteristics.

A formal power calculation has not been conducted; the planned sample of 500 patients was established based on practical considerations and the intent to obtain reasonably precise estimates of key endpoints and the recruitment capacity of participating centers. A sample of this size will allow, for example, estimation of proportions (such as adherence rate) with a sufficiently low standard error (approximately ±4-5% for proportions around 50% with a 95% confidence interval).

All statistical analyses will be performed using validated software (SPSS). A p value <0.05 will be considered indicative of statistical significance in exploratory inferential analyses.

BIBLIOGRAPHY Sillesen H, et al. Stroke Prevention by Aggressive Reduction in Cholesterol Levels Investigators. Atorvastatin reduces the risk of cardiovascular events in patients with carotid atherosclerosis: a secondary analysis of the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial. Stroke. 2008 Dec;39(12):3297-302. doi: 10.1161/STROKEAHA.108.516450.

Mach F, et al. 2025 Focused Update of the 2019 ESC/EAS Guidelines for the management of dyslipidaemias. Eur Heart J. 2025 Aug 29:ehaf190. doi: 10.1093/eurheartj/ehaf190.

Masson W, et al. LDL-C Levels Below 55 mg/dl and Risk of Hemorrhagic Stroke: A Meta-Analysis. J Stroke Cerebrovasc Dis. 2021 Apr;30(4):105655. doi: 10.1016/j.jstrokecerebrovasdis.2021.105655.

Bétrisey S, et al. Lipid-Lowering Therapy and Risk of Hemorrhagic Stroke: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2024 Feb 20;13(4):e030714. doi: 10.1161/JAHA.123.030714.

Tai SY, et al. Statin use after intracerebral hemorrhage: a 10-year nationwide cohort study. Brain Behav. 2016 May 13;6(8):e00487. doi: 10.1002/brb3.487.

Ribe AR, et al. Statins and Risk of Intracerebral Hemorrhage in Individuals With a History of Stroke. Stroke. 2020 Apr;51(4):1111-9.

ESO. Statins and ICH: ongoing controversy. Available at: https://eso-stroke.org/statins-and-ich-ongoing-controversy Rabob P, Jedsadayanmata A. Suboptimal LDL-C Goal Attainment After Ischemic Stroke and TIA: Prevalence, Determinants, and Clinical Implications. Clinics and Practice. 2025; 15(11):193.

Vandewalle L, Duchi F, Verhelle K, Vanacker P. Suboptimal lipid management in patients with acute ischemic stroke. Clin Neurol Neurosurg. 2023 Jun;229:107717.

Koenig, W., Lorenz, E.S., Beier, L. et al. Retrospective real-world analysis of adherence and persistence to lipid-lowering therapy in Germany. Clin Res Cardiol 113, 812-821 (2024).

Guglielmi V, et al. Effectiveness of adherence to lipid lowering therapy on LDL-cholesterol in patients with very high cardiovascular risk: A real-world evidence study in primary care. Atherosclerosis. 2017 Aug;263:36-41.

ELIGIBILITY:
Inclusion Criteria:

* • Recent acute cerebrovascular event, defined as a confirmed diagnosis of ischemic stroke, hemorrhagic stroke, or TIA occurring less than 30 days prior to enrollment.

  * Availability of a baseline measured LDL cholesterol value (direct or calculated) at the time of the index event or close to it.
  * Patients for whom, in routine clinical practice, a lipid-lowering therapy has been indicated and prescribed for secondary prevention (low-fat diet, supplements, statins, ezetimibe, bempedoic acid, PCSK9 inhibitors, fibrates, or other lipid-lowering agents).
  * Written informed consent obtained and signed by the patient before inclusion. If the patient is unable to provide consent autonomously (e.g., due to aphasia, impaired consciousness, etc.), informed consent will be obtained from a legal representative or proxy, in accordance with applicable regulations.

Exclusion Criteria:

* • Comorbidities or conditions preventing 3-month follow-up: e.g., terminal oncological disease with life expectancy <3 months, severe cognitive impairment (e.g., advanced dementia), or other conditions that make it impossible to obtain follow-up information; inability to contact the patient after discharge (e.g., non-resident foreign patient or lacking telephone contacts).

  * Any other clinical, psychological, or social condition that, in the investigator's judgment, may compromise the patient's ability to adhere to the study or the reliability of the collected data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included with any etiological subtype of ischemic stroke (e.g., cardioembolic, atherosclerotic, lacunar, etc.) or hemorrhagic stroke or TIA.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to lipid-lowering therapy | 3 months
  Adherence to lipid-lowering therapy, defined as the percentage of patients who are adherent (intake of ≥80% of prescribed doses) and persistent (on therapy without interruptions) at the end of follow-up. Rates of persistence (patients who did not discontinue therapy) and adherence (patients who took it regularly) may also be considered separately.

SECONDARY OUTCOMES:
Proportion of patients achieving an LDL target value | 3 months
  Proportion of patients achieving an LDL target value (for example, <55 mg/dL for ischemic stroke patients, <40 mg/dL for patients already on maximal therapy, etc.) at the 90 ± 15-day follow-up. This endpoint reflects the overall effectiveness of lipid-lowering management in bringing patients to the recommended target.
Recurrence of stroke (ischemic or hemorrhagic), TIA, or acute cardiovascular events | 3 months
  Recurrence of stroke (ischemic or hemorrhagic), TIA, or acute cardiovascular events (myocardial infarction or angina) within 90 ± 15 days of the index event (composite endpoint). The incidence of recurrent ischemic stroke, hemorrhagic stroke, and TIA will also be analyzed separately as secondary individual endpoints.
All-cause mortality | 3 months
  All-cause mortality at 90 ± 15 days. In parallel, cerebrovascular mortality (deaths attributable to the direct consequences of stroke or other cerebrovascular events) will be analyzed relative to mortality from other causes.
Adverse events related to lipid-lowering medications | 3 months
  Adverse events related to lipid-lowering medications: incidence of clinically relevant side effects reported within 90 ± 15 days (e.g., myalgias without significant CK elevation, gastrointestinal disturbances from fibrates, injection-site reactions with PCSK9 inhibitors, etc.). These will contribute to the overall evaluation of therapy tolerability.
Functional disability | 3 months
  Functional disability at 90 ± 15 days: optionally assessed using the mRS (modified Rankin Scale) score if captured at follow-up, to provide an overview of overall clinical outcome.

IPD SHARING:
Plan to Share IPD: Undecided